CLINICAL TRIAL: NCT05464901
Title: The Real-World Treatment Status of Venous Thromboembolism and the Related Factors Associated With Higher Rates of PE After a DVT in Southwestern China
Brief Title: VTE and the Related Factors Associated With Higher Rates of PE After a DVT in Southwestern China
Status: Completed | Type: Observational
Sponsor: Wei Huang (Other)
Responsible Party: Sponsor-Investigator, Wei Huang, Professor, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: 2019XMSB0005627
Record Dates: First submitted 2022-07-15; First posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Venous Thromboembolism; Deep Vein Thrombosis; Pulmonary Embolism; Anticoagulants
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Little is known about the current management status of venous thromboembolism (VTE) in Southwestern China. We aimed to investigate the status of anticoagulant administration in VTE in Southwestern China and assess the potential predictors of deep vein thrombosis (DVT) complicated pulmonary embolism (PE). We extracted data from YiduCloud database from December 2006 to November 2018 and performed a cross-sectional survey of VTE. The demographics, laboratory tests, and anticoagulants were collected and analyzed in the logistic regression model, classification tree and Random Forest model.

DETAILED DESCRIPTION:
We established a collaborative epidemiological work of southwestern China for our cross-sectional survey sample, which included hospitalized patients in the seven main medical centers who met the inclusion criteria. The Human Research Committee of Chongqing Medical University approved this study and waived the need for informed consent. Patients were eligible to be included in the study if they are admitted or discharged with a diagnosis of DVT or/and PE and if they ever received treatment in the seven medical centers between December 2006 to November 2018.

ELIGIBILITY:
Inclusion Criteria:

- In the Chinese VTE guidelines, the diagnosis of VTE depends on a series of tests. D-dimer was used to screen for thrombosis, and limb venous ultrasound was used to diagnose DVT. CT pulmonary angiography (CTPA) or pulmonary ventilation perfusion scan was used for the diagnosis of pulmonary embolism. Through the retrieval of patient diagnosis in the database, we retrieved the basic data of all patients diagnosed as VTE during the study period.

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: In the patients' characteristics, the hypertensive disorders of pregnancy were defined and classified into (a) hypertension known before pregnancy or present in the first 20 weeks and (b) hypertension arising de novo at or after 20 weeks on the basis of the International Society for the Study of Hypertension in Pregnancy Classification, Diagnosis, and Management Recommendations for International Practice
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2006-12-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
The maternal cardiac events and the neonatal complications | 2010-2019
  Primary outcomes of interest were major adverse cardiac events (MACEs), obstetric complications and neonatal adverse clinical events (NACEs).

IPD SHARING:
Plan to Share IPD: Undecided